CLINICAL TRIAL: NCT04368936
Title: Relationship Between Polymorphisms of TRPV1 and KCC2 Gene in Children With Febrile Seizures
Status: Completed | Type: Observational
Sponsor: Institut za Rehabilitaciju Sokobanjska Beograd (Other)
Responsible Party: Principal Investigator, Tamara Filipovic, Principal Investigator, Institut za Rehabilitaciju Sokobanjska Beograd
Other Study IDs: SBCPRN2
Record Dates: First submitted 2020-04-24; First posted 2020-04-30 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Febrile Seizure
Keywords: gene polymorphisms; febrile seizure; KCC2 gene; TRPV1 gene
MeSH Terms: conditions — Seizures, Febrile | interventions — Real-Time Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — * C_16186074_10 for rs2297201 polymorphisms KCC2 gene
  * C_1093688_20 za rs222747 polymorphisms TRPV1 gene (Thermo Fisher Scientific, Walthman, MA, SAD)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- FS: Febrile Seizures: Involved patient with diagnosed Febrile Seizures which were hospitalized or recieved ambulatory treatment in University Children´s Hospital in Belgrade. Ages 1-14 years
  Interventions: Genetic: Isolated DNA, Real Time PCR
- CN: Control group: The control group was made of healthy children older than 5 years of age, which have never had any neurological disorders in their anamnesis and who were patients in preschool or school dispensaries in the city of Belgrade
  Interventions: Genetic: Isolated DNA, Real Time PCR
- SFS : group of individuals with simple FS: Simplex febrile seizures (SFS) last shorter than 15 minutes and their type is tonic-clonic. Also, they did not show signs of recidivism during the first 24 hours and were diagnosed at the patients aged from 6th months to 5th year
  Interventions: Genetic: Isolated DNA, Real Time PCR
- CFS : group of individuals with complex FS: Complex febrile seizures (CFS) were diagnosed at those patients that had focal seizure or epileptic status or seizure having the body temperature lower than 38 degree, which occurred outside of the typical age group and finally which repeated in the first 24 hours again
  Interventions: Genetic: Isolated DNA, Real Time PCR
- WFS: group of individuals with FS and without epilepsia: group of children with Febrile Seizure and not developed Epilepsia
  Interventions: Genetic: Isolated DNA, Real Time PCR
- EFS: group of individuals with Epilepsia and Febrile Seizures: Group of children with Febrile Seizures, who have developed Epilepsy
  Interventions: Genetic: Isolated DNA, Real Time PCR

INTERVENTIONS:
Genetic: Isolated DNA, Real Time PCR — We are isolated DNA from the blood sample. To determine the genotypes of the analyzed polymorphisms use real-time PCR using TaqMan essays.
  When analyzing the KCC2 polymorphisms, the VIC dye gene corresponded to the C allele, and the FAM dye corresponded to the T allele, while at the TRPV1 gene polymorphism, the VIC dye corresponded to the C allele and the FAM dye to the G allele.

SUMMARY:
Febrile seizures (FS) are the most common neurological disorder in chilhood. The etiology of FN is still the subject of numerous studies and it is known that it can depend on genetic predisposition.

DETAILED DESCRIPTION:
Febrile seizures (FS) are the most common neurological disorder in chilhood. It is precisely because of the high incidence of the disease, the age that includes the tendency of repetition, represent a particular challenge in pediatric practice.

FS, as defined by the American Academy of Pediatrics (AAP), are " seizure occurring in febrile children between the ages of 6 and 60 months who do not have an intracranial infection, metabolic disturbance, or history of afebrile seizures ".

Simple febrile seizure is defined as a short (<15 min) generalized seizure, not repeat within 24 h, that occurs during a febrile illness not resulting from an acute disease of the nervous system in a child aged between 6 months and 5 years, with no neurologic deficits and no previous afebrile seizures. Complex febrile seizures are a focal, or generalized and prolonged seizure, of a duration of greater than 15 min, recurring more than once in 24 h, and/or associated with postictal neurologic abnormalities, more frequently a postictal palsy (Todd's palsy), or with previous neurologic deficits.

The etiology of FN is still the subject of numerous studies and it is known that it can depend on genetic predisposition.

Animal studies have shown that mice without the KCC2 gene have frequent generalized seizures, while those with heterozygous deletion of the KCC2 gene have a reduced threshold for seizure onset. In the human population, mutations of this gene have been reported in children with FN as well as in children with epilepsy. There is no examined an association between polymorphism rs2297201 KCC2 gene and FS.

Studies have shown an association between TRPV1 genes and the appearance of FS in experimental models, however, similar studies in the human population have not been done so far. Studies Moria et al. 2012 showed that polymorphism rs222797 TRPV1 gene involve the regulation of human cortical excitability, glutamate transmission and increased neuronal excitability. The C allele this polymorphism is associated with a greater maximal response to the caspaicin and anadamine agonists. All of this indicate that changes TRPV1 gene that lead to increased channel function may suggest a predisposition for FS.

Since FS are genetically controlled, we want to determine the association of TRPV1 and KCC2 gene polymorphisms with the occurrence of FN.

ELIGIBILITY:
Inclusion Criteria:

* Our research involve patient with diagnosed Febrile Seizure which were hospitalized or recieved ambulatory treatment in University Children´s Hospital in Belgrade
* For each patient, a diagnosis of FS was made based on the ILAE definition (International Leage
* The main criterion for inclusion in the study was enhanced FS without prior occurrence of afebrile seizure.

Exclusion Criteria:

* Patients with evidence of intracranial infections and metabolic disbalance
* Patients with incomplited medical documentation

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The Febrile Seizure affected children as well as the individuals from the control group were members of the same population (Serbian).
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Detection of the polymorphism in the TRPV1 gene polymorphisms | 2 weeks
  The detection of the polymorphism in the TRPV1 gene will be done by the PCR Real time method: During PCR ampification, in addition to primers, an allele of specific oligonucleotide probes is used, which at the 5 'end is labeled with specific fluorescent dye (Reporter dye, eg VIC and FAM), while at the 3' position there is a quencher, which is the role of blocking fluorescence emissions.The fluorescence intensity increases during each cycle and allows us to monitor dynamic reactions in real time.After the final PCR reaction, increasing the fluorescence of the dyes is displayed on the heterozygosity of the test allele. Fluorescence coupling of only one color indicates a homozygous state.VIC dye corresponds to allele C, and FAM dye to allele G.
Detection of the polymorphism in the KCC2 gene polymorphisms | 2 weeks
  The detection of the polymorphism in the KCC2 gene will be done by the PCR Real time method: During PCR ampification, in addition to primers, an allele of specific oligonucleotide probes is used, which at the 5 'end is labeled with specific fluorescent dye (Reporter dye, eg VIC and FAM), while at the 3' position there is a quencher, which is the role of blocking fluorescence emissions.The fluorescence intensity increases during each cycle and allows us to monitor dynamic reactions in real time.After the final PCR reaction, increasing the fluorescence of the dyes is displayed on the heterozygosity of the test allele. Fluorescence coupling of only one color indicates a homozygous state. VIC dye corresponds to allele C, and FAM dye to allele T.

CONTACTS AND LOCATIONS:
Overall Officials: Sanja Dimitrijevic, PhD, Principal Investigator — Specila hospital for cerebral palsy and developmental neurology

IPD SHARING:
Plan to Share IPD: Yes
All of individual participant data collected during the trial, after deindetification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately after publication. No end date.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Background] Leung AK, Hon KL, Leung TN. Febrile seizures: an overview. Drugs Context. 2018 Jul 16;7:212536. doi: 10.7573/dic.212536. eCollection 2018. PMID 30038660
- [Background] Dimitrijevic S, Cvjeticanin S, Pusica A, Jekic B, Filipovic T, Nikolic D. Anthropogenetic Variability in the Group of Individuals with Febrile Seizures: Population-Genetic Study. Biomed Res Int. 2018 Jul 5;2018:7845904. doi: 10.1155/2018/7845904. eCollection 2018. PMID 30069480
- [Background] Reid AY, Riazi K, Campbell Teskey G, Pittman QJ. Increased excitability and molecular changes in adult rats after a febrile seizure. Epilepsia. 2013 Apr;54(4):e45-8. doi: 10.1111/epi.12061. Epub 2013 Jan 7. PMID 23293960
- [Background] Puskarjov M, Seja P, Heron SE, Williams TC, Ahmad F, Iona X, Oliver KL, Grinton BE, Vutskits L, Scheffer IE, Petrou S, Blaesse P, Dibbens LM, Berkovic SF, Kaila K. A variant of KCC2 from patients with febrile seizures impairs neuronal Cl- extrusion and dendritic spine formation. EMBO Rep. 2014 Jun;15(6):723-9. doi: 10.1002/embr.201438749. Epub 2014 Mar 24. PMID 24668262
- [Background] Huang WX, Yu F, Sanchez RM, Liu YQ, Min JW, Hu JJ, Bsoul NB, Han S, Yin J, Liu WH, He XH, Peng BW. TRPV1 promotes repetitive febrile seizures by pro-inflammatory cytokines in immature brain. Brain Behav Immun. 2015 Aug;48:68-77. doi: 10.1016/j.bbi.2015.01.017. Epub 2015 Mar 20. PMID 25801060
- [Background] Xu H, Tian W, Fu Y, Oyama TT, Anderson S, Cohen DM. Functional effects of nonsynonymous polymorphisms in the human TRPV1 gene. Am J Physiol Renal Physiol. 2007 Dec;293(6):F1865-76. doi: 10.1152/ajprenal.00347.2007. Epub 2007 Oct 3. PMID 17913835